CLINICAL TRIAL: NCT04305483
Title: Evaluation of the Color Change of the Laser and Chemical Vital Whitening Method in the Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Beyza Ünalan Değirmenci, Assistant Professor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 05.12.2013/07
Record Dates: First submitted 2020-03-08; First posted 2020-03-12 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Color; Change Teeth, Posteruptive
Keywords: Vital Bleaching; Color measurement; spectrophotometer

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser Bleaching (Active Comparator): 35% Hydrogen peroxide, potassium nitrate, sodium fluoride, sodium hydroxide, thickener, glycol derivative containing bleaching agent activated with diode laser
  Interventions: Procedure: Laser Bleaching
- Chemical Bleaching (Active Comparator): 35% Hydrogen peroxide, thickener, plant extracts, amide, release agent, glycol, paint and water containing chemical bleaching agent used for control group without a laser activation
  Interventions: Procedure: Chemical Bleaching

INTERVENTIONS:
Procedure: Laser Bleaching — Content; There are 35% hydrogen peroxide, potassium nitrate, sodium fluoride, sodium hydroxide, thickener, glycol derivative. The way of application; Gingival protection is applied. The gel is applied to the labial surfaces of the teeth with a thickness of 1-2 mm. The use of laser increases the effectiveness of the gel. Operator and patient use protective glasses during laser application. The gel shows its effectiveness in about eight minutes. Then the gel is removed with the help of saliva absorber. The procedure is repeated until the desired degree of whitening is achieved. Then it is checked with a color scale.
  Arms: Laser Bleaching
Procedure: Chemical Bleaching — "Total Blanc Office Teeth Whitening System (H35)" will be used as chemical whitening agent. Content; There are 35% hydrogen peroxide, thickener, plant extracts, amide, release agent, glycol, paint and water. Method of Application; Gingival protection is applied. A 1 mm thick layer of gel is applied to all of the labial surfaces of the tooth. The whitening agent remains on the tooth surface for 20 minutes. At the end of this period, the gel is removed with saliva absorber and the surface is cleaned with a moist gauze.
  Arms: Chemical Bleaching

SUMMARY:
Having an aesthetic smile has become very common among patients today. Recent studies have shown that people aged 18-49 want to have whiter and brighter teeth. The demand for whitening has increased by 300% in the last 5 years. New materials and equipment have been developed to meet this demand, and various whitening techniques have been developed for use at home and in clinical practice. Determination of color in dentistry; It can be divided into two categories with the help of visual and computer-aided devices. Eye color determination is the most widely used method during the construction of a indirect restoration. The evaluation of tooth color by eye is quite subjective. Physiological variables such as external light source, experience, age and human eye fatigue, color blindness cause inadequate results. Due to interpersonal detection differences during color perception, the lack of standardization in the determination of tooth color can be improved with the use of computer-aided devices such as spectroradiometer, spectrophotometer, colorimeter and with the help of film-based photographs and digital photographs. Spectrophotometric approach; the point of view is interesting, as it allows for an objective application, regardless of the practitioner's experience. The color selection made with the use of these devices provides a potential advantage over the color selection made with the eye. Because these measurements are objective, can be counted and can be obtained faster. Although widespread uses of computer aided colorimeters and spectrophotometers have been reported in dental studies, most devices are not suitable for routine clinical use. Color analysis with these computer-aided devices may cause inaccurate results especially in the evaluation of translucent objects such as teeth. Therefore, a combination using both eyes and devices should be used.

DETAILED DESCRIPTION:
Tooth color; It is formed by the combination of enamel, dentin and pulp with different optical properties. Tooth coloring is divided into two as etiological, internal and external. External colorants can be removed simply by cleaning. Removal of intrinsic coloring is possible with chemical bleaching. In the treatment of tooth coloring, whitening is considered the least aggressive method.

Due to the increasing interest in aesthetics in recent years, patients' demands for teeth whitening have increased. Home-bleaching technique, developed by Haywood and Heymann in 1989, has been the most frequently used method until recently. In this method, the bleaching agent contains 10% hydrogen peroxide. For 2-5 weeks, whitening is performed by placing the gel in a plate by the patient every night. The advantages of this method are that it is easy to apply, low cost, use of lower rates of hydrogen peroxide, and less time spent in the clinic. However, the disadvantages are that the whitening process is not under the control of the physician, the patient does not apply the whitening gel regularly, and the procedure takes several weeks. Office-bleaching technique has been developed in order to make the bleaching process more controlled, to ensure color stability and to shorten the time. This technique, which contains a high concentration of (15-38%) hydrogen peroxide, is activated by heat or light sources. These sources include plasma arc, LED, UV lamps and laser. However, there is no consensus on the effectiveness of heat and light sources used in tooth whitening.

The light sources used during bleaching are expected to increase the effectiveness of the bleaching and shorten the processing time. Among these, plasma arc and diode lasers have a wide range of uses. Laser teeth whitening method has been applied for about 15 years and many laser devices have been recommended for this procedure. It is expected that the treatment time will decrease and the sensitivity that may occur in the teeth will decrease as a result of laser application. However, the superiority of laser bleaching compared to other methods is still controversial.

External root resorption and irritation in soft tissues can be observed during the teeth whitening, even if in a small amount. It is stated that the sensitivity of teeth after the procedure is the most common complication by some researchers, but disappears by itself after the end of the bleaching process.

The purpose of aesthetic applications in dentistry; morphological, optical and biological compatibility. Tooth color is one of the most important criteria of aesthetics. Clinically, two different methods are used in color selection. The first, visual method, includes evaluation with the naked eye. The second method is colorimeter, spectrophotometer etc. is the use of devices that measure color. During clinical applications, color selection of dental materials is done by using visual scales. Color selection by visual method is both subjective and difficult; it can also lead to inadequate results. During color selection, erroneous results may occur due to parameters such as ambient light, physician's experience and age, and eye fatigue.

Due to these existing disadvantages, systems such as spectrophotometers, colorimeters, digital color meters have been launched to assist the physician in color selection. In dentistry, spectrophotometers and colorimeters are used to overcome problems related to color selection with the eye. Although the visual method is used more in the selection of colors by clinicians, it is stated that the color measurements made by using the visual method and spectrophotometer together are quite successful.

Color is formed by the merge of wavelengths in a light beam. In order for an object to be visible, it must emit light or reflect light from a light source. From the point of view of dentistry, the property of objects to reflect the incoming light is more important. The incoming light usually consists of a mixture of various wavelengths, that is, it has a polychromatic feature. When light comes on an object, it absorbs certain wavelengths and reflects certain wavelengths. The human eye can distinguish light between wavelengths of 400-700 nμ. Nerve responses play a big role in the appearance of color. As a result of attached stimulation, the eye gets tired and the reaction of the eye decreases. Color separation is a subjective issue.

The first color specification was proposed by CIE in 1931. Although this system was developed in the following years, its principles have still not changed. CIE system uses 3 variables, X, Y and Z. These variables are based on the spectral response functions defined by the CIE observer. The CIE chromaticity diagram is also used to define the exact color. In another CIE color system, three variables are used: L *, a * and b *.

The spectrophotometer is a photometric appliance that is used to measure the transmittance, reflection and true absorption of color. They contain prisms or dispersing parts to create a continuous color line in their structure. Spectrophotometric color measurements may vary depending on the light source used and the measurement mode. Some spectrophotometers can be used according to two different measurement modes: Specular Component Included (SCI) and Excluded (SCE). Many types of standard light source are also used for color measurement of dental materials. These devices give three stimulus values x, y, z or CIE L *, a *, b *. These values can be converted into numerical values and color variables of different objects can be compared.

The aim of the study is to compare the color change caused by laser-activated and chemically activated vital whitening systems with two different evaluation methods (digital camera and spectrophotometer). In this way, a comparison of the effectiveness of both the whitening systems and the reliability of the evaluation methods will be made. It is also aimed to determine the sensitivity of the teeth that may occur during and after bleaching.

ELIGIBILITY:
Inclusion Criteria:

1. Systemically healthy individuals
2. Non-smokers
3. Those who do not consume more than three cups of tea / coffee per day
4. No devital and / or restorated teeth in the upper anterior six teeth

Exclusion Criteria:

1. Pregnancy
2. Patient with hypersensitivity
3. Patient with crack, exposed dentin
4. Patients with dental caries
5. Patient who have gingival recession

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-12-01 (Actual); Primary Completion 2014-02-24 (Actual); Study Completion 2014-03-13 (Actual)

PRIMARY OUTCOMES:
Color change according to CIE Lab system | Immediately after procedure
  Before and after the bleaching procedure color of the maxillary anterior teeth were measured based on CIE Lab system with a spectrophotometer and digital photography machine.
Color change according to CIE Lab system | After 2 weeks
  Before and after the bleaching procedure color of the maxillary anterior teeth were measured based on CIE Lab system with a spectrophotometer and digital photography machine.

SECONDARY OUTCOMES:
Evaluation of the Procedural Sensitivity Levels | Immediately after procedure
  After the related bleaching procedure, operator wanted to evaluate sensitivity levels of the patients according to visual analogue scale.
Evaluation of the Procedural Sensitivity Levels | After 2 weeks
  After the related bleaching procedure, operator wanted to evaluate sensitivity levels of the patients according to visual analogue scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Beyza Ünalan Değirmenci, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hahn P, Schondelmaier N, Wolkewitz M, Altenburger MJ, Polydorou O. Efficacy of tooth bleaching with and without light activation and its effect on the pulp temperature: an in vitro study. Odontology. 2013 Jan;101(1):67-74. doi: 10.1007/s10266-012-0063-4. Epub 2012 Mar 1. PMID 22395767
- [Result] Kivanc BH, Arisu HD, Ulusoy OI, Saglam BC, Gorgul G. Effect of light-activated bleaching on pulp chamber temperature rise: an in vitro study. Aust Endod J. 2012 Aug;38(2):76-9. doi: 10.1111/j.1747-4477.2010.00271.x. Epub 2010 Oct 24. PMID 22827820
- [Result] Lima DA, Aguiar FH, Liporoni PC, Munin E, Ambrosano GM, Lovadino JR. In vitro evaluation of the effectiveness of bleaching agents activated by different light sources. J Prosthodont. 2009 Apr;18(3):249-54. doi: 10.1111/j.1532-849X.2008.00420.x. Epub 2009 Feb 2. PMID 19210610